CLINICAL TRIAL: NCT01973569
Title: A Confirmatory Study of AMG 162 (Denosumab) in Patients With Rheumatoid Arthritis on DMARDs Treatment (Phase III)
Brief Title: AMG 162 (Denosumab) Phase 3 Study (DESIRABLE Study) in Participants With Rheumatoid Arthritis on Disease-modifying Antirheumatic Drugs (DMARDs) Treatment
Acronym: DESIRABLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMG162-D-J301
Record Dates: First submitted 2013-10-25; First posted 2013-10-31 (Estimated); Results first posted 2019-12-13 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Denosumab; RANKL; RANK; AMG 162; joint damage; Developmental Phase III
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Denosumab 6 months (Experimental): denosumab administered subcutaneously every 6 months
  Interventions: Drug: denosumab
- Denosumab 3 months (Experimental): denosumab administered subcutaneously every 3 months
  Interventions: Drug: denosumab
- placebo (Placebo Comparator): placebo administered subcutaneously to match denosumab
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: denosumab — denosumab administered subcutaneously
  Other Names: AMG 162
  Arms: Denosumab 3 months; Denosumab 6 months
Drug: placebo — placebo administered subcutaneously to match denosumab
  Arms: placebo

SUMMARY:
To evaluate the inhibitory effect of progression, compared with placebo, in joint destruction by AMG 162 administered subcutaneously to rheumatoid arthritis participants.

DETAILED DESCRIPTION:
To evaluate the inhibitory effect of progression, compared with placebo, in joint destruction by AMG 162 administered subcutaneously at a dose of 60 mg every 6 months or every 3 months for 12 months to rheumatoid arthritis participants.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with rheumatoid arthritis according to the American College of Rheumatology (ACR) criteria for rheumatoid arthritis classification (1987 revision) or the 2010 ACR-EULAR (The European League Against Rheumatism) classification criteria for rheumatoid arthritis

Exclusion Criteria:

* Functional class IV according by the ACR revised classification (1991)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 679 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2017-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tsutomu Takeuchi, Prof., Study Director — Division of Rheumatology Department of Internal Medicine, Keio University
Locations (1):
- Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https:// vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Tanaka Y, Takeuchi T, Soen S, Yamanaka H, Yoneda T, Tanaka S, Nitta T, Okubo N, Genant HK, van der Heijde D. Effects of Denosumab in Japanese Patients With Rheumatoid Arthritis Treated With Conventional Antirheumatic Drugs: 36-month Extension of a Phase III Study. J Rheumatol. 2021 Nov;48(11):1663-1671. doi: 10.3899/jrheum.201376. Epub 2021 Apr 15. PMID 33858976
- [Derived] Takeuchi T, Soen S, Ishiguro N, Yamanaka H, Tanaka S, Kobayashi M, Okubo N, Nitta T, Tanaka Y. Predictors of new bone erosion in rheumatoid arthritis patients receiving conventional synthetic disease-modifying antirheumatic drugs: Analysis of data from the DRIVE and DESIRABLE studies. Mod Rheumatol. 2021 Jan;31(1):34-41. doi: 10.1080/14397595.2019.1703484. Epub 2020 Jan 9. PMID 31826682

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 679 participants who met all inclusion and none of the exclusion criteria were included in the study; efficacy outcomes were assessed in the Full Analysis Set (n=654).
Period: Overall Study
Arm/Group | Denosumab 6 Months | Denosumab 3 Months | Placebo
Started | 228 | 225 | 226
Received Study Drug | 222 | 222 | 223
Did Not Receive Study Drug | 6 | 3 | 3
Discontinued Study Treatment | 23 | 22 | 15
Discontinued Study | 23 | 22 | 15
Completed | 199 | 200 | 208
Not Completed | 29 | 25 | 18
Not completed — Adverse Event | 9 | 2 | 4
Not completed — Protocol Violation | 2 | 1 | 3
Not completed — Withdrawal by Subject | 7 | 5 | 2
Not completed — Invasive dental treatment | 3 | 5 | 6
Not completed — Prohibited concomitant d | 1 | 5 | 0
Not completed — Disease progression | 0 | 3 | 0
Not completed — Other | 1 | 1 | 0
Not completed — Did not receive study drug | 6 | 3 | 3

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis Population included participants in the Full Analysis Set (FAS). The FAS was defined as all randomized participants excluding those who met any of the following criteria:
  * Received no investigational product
  * Had no baseline TSS or no available TSS after the first administration of the investigational product
Groups:
- Total: Total of all reporting groups
Arm/Group | Denosumab 6 Months | Denosumab 3 Months | Placebo | Total
Number analyzed (Participants) | 217 | 219 | 218 | 654
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 140 | 150 | 163 | 453
  >=65 years | 77 | 69 | 55 | 201
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (12.3) | 58.2 (12.04) | 55.8 (11.7) | 57.4 (12.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 168 | 154 | 167 | 489
  Male | 49 | 65 | 51 | 165
Region of Enrollment [Number; unit: participants]
  Japan | 217 | 219 | 218 | 654
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 22.38 (3.68) | 22.64 (3.62) | 22.65 (3.49) | 22.56 (3.59)

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Sharp Score (TSS) From Baseline to Month 12 Following Subcutaneous Administration of Denosumab or Placebo
Description: Change from baseline in Total Sharp Score (TSS) from baseline to month 12 was assessed. The TSS was defined as the sum of the erosion score and the joint space narrowing scores from radiographic assessments. The maximum radiographic TSS from the both hands/wrists and both feet is 448. Higher values represented greater damage.
Time Frame: baseline to month 12
Population: TSS was assessed in Full Analysis Set.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Denosumab 6 Months | Denosumab 3 Months | Placebo
Number analyzed (Participants) | 217 | 219 | 218
score on a scale | 0.99 [0.49 to 1.49] | 0.72 [0.41 to 1.03] | 1.49 [0.99 to 1.99]
Statistical Analysis 1: Comparison: Denosumab 6 Months vs Placebo; Test type: Superiority; p = 0.0235, van Elteren stratified rank test — The hierarchical testing procedure was applied for multiple comparisons of the primary endpoint. First, comparison between AMG 162 60mg Q3M vs placebo is tested. Only if it is rejected, comparison of AMG 162 60mg Q6M vs placebo is formally tested; van Elteren stratified rank test adjusting for baseline use of glucocorticoid was used

2. Secondary Outcome: Change in Total Sharp Score (TSS) From Baseline to Month 6 Following Subcutaneous Administration of Denosumab or Placebo
Description: Change from baseline in Total Sharp Score (TSS) from baseline to month 6 was assessed. The TSS was defined as the sum of the erosion score and the joint space narrowing scores from radiographic assessments. The maximum radiographic TSS from the both hands/wrists and both feet is 448. Higher values represented greater damage.
Time Frame: baseline to month 6
Population: TSS was assessed in the Full Analysis Set.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Denosumab 6 Months | Denosumab 3 Months | Placebo
Number analyzed (Participants) | 217 | 219 | 218
score on a scale | 0.62 [0.27 to 0.98] | 0.48 [0.24 to 0.72] | 0.92 [0.60 to 1.23]
Statistical Analysis 1: Comparison: Denosumab 6 Months vs Placebo; Test type: Superiority; p = 0.0360, van Elteren stratified rank test; van Elteren stratified rank test adjusting for baseline use of glucocorticoid was used

3. Secondary Outcome: Change in Erosion Score From Baseline to Month 6 Following Subcutaneous Administration of Denosumab or Placebo
Description: Change from baseline in Erosion Score from baseline to month 6 was assessed. The Erosion Score was defined for the sum of the joint level erosion scores among the 44 joints in both hands/wrist and both feet from radiographic assessments using the van der Heijde modified Sharp scoring method. The maximum radiographic Erosion Score from both hands/wrist and both feet is 280. Higher values represented greater damage.
Time Frame: baseline to month 6
Population: The Erosion Score was assessed in the Full Analysis Set.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Denosumab 6 Months | Denosumab 3 Months | Placebo
Number analyzed (Participants) | 217 | 219 | 218
score on a scale | 0.34 [0.16 to 0.53] | 0.13 [0.03 to 0.24] | 0.58 [0.39 to 0.78]
Statistical Analysis 1: Comparison: Denosumab 6 Months vs Placebo; Test type: Superiority; p = 0.1323, van Elteren stratified rank test; van Elteren stratified rank test adjusting for baseline use of glucocorticoid was used

4. Secondary Outcome: Change in Joint Space Narrowing From Baseline to Month 6 Following Subcutaneous Administration of Denosumab or Placebo
Description: Change from baseline in Joint Space Narrowing from baseline to month 6 was assessed. Joint Space Narrowing was defined for the sum of the joint level joint space narrowing scores among the 42 joints in both hands/wrist and both feet from radiographic assessments using the van der Heijde modified Sharp scoring method. The maximum radiographic Joint Space Narrowing from both hands/wrists and both feet is 168. Higher values represented greater damage.
Time Frame: baseline to month 6
Population: Joint Space Narrowing was assessed in the Full Analysis Set.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Denosumab 6 Months | Denosumab 3 Months | Placebo
Number analyzed (Participants) | 217 | 219 | 218
score on a scale | 0.28 [0.07 to 0.50] | 0.35 [0.17 to 0.53] | 0.33 [0.18 to 0.48]
Statistical Analysis 1: Comparison: Denosumab 6 Months vs Placebo; Test type: Superiority; p = 0.0448, van Elteren stratified rank test; van Elteren stratified rank test adjusting for baseline use of glucocorticoid was used

5. Secondary Outcome: Change in Erosion Score From Baseline to Month 12 Following Subcutaneous Administration of Denosumab or Placebo
Description: Change from baseline in Erosion Score from baseline to month 12 was assessed. The Erosion Score was defined for the sum of the joint level erosion scores among the 44 joints in both hands/wrist and both feet from radiographic assessments using the van der Heijde modified Sharp scoring method. The maximum radiographic Erosion Score from both hands/wrist and both feet is 280. Higher values represented greater damage.
Time Frame: baseline to month 12
Population: The Erosion Score was assessed in the Full Analysis Set.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Denosumab 6 Months | Denosumab 3 Months | Placebo
Number analyzed (Participants) | 217 | 219 | 218
score on a scale | 0.51 [0.22 to 0.80] | 0.22 [0.09 to 0.34] | 0.98 [0.65 to 1.31]
Statistical Analysis 1: Comparison: Denosumab 6 Months vs Placebo; Test type: Superiority; p = 0.0104, van Elteren stratified rank test; van Elteren stratified rank test adjusting for baseline use of glucocorticoid was used

6. Secondary Outcome: Change in Joint Space Narrowing From Baseline to Month 12 Following Subcutaneous Administration of Denosumab or Placebo
Description: Change from baseline in Joint Space Narrowing from baseline to month 12 was assessed. Joint Space Narrowing was defined for the sum of the joint level joint space narrowing scores among the 42 joints in both hands/wrist and both feet from radiographic assessments using the van der Heijde modified Sharp scoring method. The maximum radiographic Joint Space Narrowing from both hands/wrists and both feet is 168. Higher values represented greater damage.
Time Frame: baseline to month 12
Population: Joint Space Narrowing was assessed in the Full Analysis Set.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Denosumab 6 Months | Denosumab 3 Months | Placebo
Number analyzed (Participants) | 217 | 219 | 218
score on a scale | 0.48 [0.20 to 0.76] | 0.50 [0.27 to 0.74] | 0.51 [0.28 to 0.74]
Statistical Analysis 1: Comparison: Denosumab 6 Months vs Placebo; Test type: Superiority; p = 0.2570, van Elteren stratified rank test; van Elteren stratified rank test adjusting for baseline use of glucocorticoid was used

7. Secondary Outcome: Percent Change in Bone Mineral Density (BMD) From Baseline to Month 12 Following Subcutaneous Administration of Denosumab or Placebo
Description: The percent change from baseline in Bone Mineral Density (BMD) to month 12 was assessed. Bone mineral density (BMD) was measured by dual x-ray absorptiometry (DXA).
Time Frame: baseline to month 12
Population: Bone mineral density was assessed in the Full Analysis Set.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Denosumab 6 Months | Denosumab 3 Months | Placebo
Number analyzed (Participants) | 217 | 219 | 218
percent change | 3.99 (0.24) | 4.88 (0.24) | -1.03 (0.25)
Statistical Analysis 1: Comparison: Denosumab 6 Months vs Placebo; Test type: Superiority; p < 0.0001, Regression, Cox; ANCOVA model adjusting for treatment, baseline (BL) value, machine type, BL value-by-machine type interaction, and BL use of glucocorticoid was used; Mean Difference (Net) = 5.02, 95% CI 2-sided [4.41 to 5.63]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the first dose to the last dose of study drug, up to 12 months.
Description: Adverse events that emerge (or worsen) from the first dose of study drug to the last dose of study drug were reported in the Safety Analysis Set. The Safety Analysis Set was defined as all enrolled participants who received at least one dose of the investigational product. One participant of the Denosumab 6 months group was administered the placebo mistakenly, and was thus included in the placebo group for the safety analysis.
Arm/Group | Denosumab 6 Months | Denosumab 3 Months | Placebo
All-Cause Mortality (participants affected / at risk) | 0/221 | 1/222 | 0/224
Serious Adverse Events (participants affected / at risk) | 19/221 | 19/222 | 13/224
Other Adverse Events (participants affected / at risk) | 127/221 | 122/222 | 125/224
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Denosumab 6 Months (N=221) | Denosumab 3 Months (N=222) | Placebo (N=224)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0 | 0
Paroxysmal arrhythmia (Cardiac disorders) | 0 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Spinal muscular atrophy (Congenital, familial and genetic disorders) | 0 | 1 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 1
Mass (General disorders) | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Abscess jaw (Infections and infestations) | 1 | 0 | 0
Arthritis bacterial (Infections and infestations) | 0 | 1 | 0
Atypical mycobacterial infection (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Tuberculosis (Infections and infestations) | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Brain stem infarction (Nervous system disorders) | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0
Device dislocation (Product Issues) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0
Calculus bladder (Renal and urinary disorders) | 1 | 0 | 0
Prerenal failure (Renal and urinary disorders) | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Denosumab 6 Months (N=221) | Denosumab 3 Months (N=222) | Placebo (N=224)
Dental caries (Gastrointestinal disorders) | 12 | 7 | 9
Stomatitis (Gastrointestinal disorders) | 22 | 27 | 13
Hepatic function abnormal (Hepatobiliary disorders) | 14 | 13 | 20
Influenza (Infections and infestations) | 8 | 10 | 12
Nasopharyngitis (Infections and infestations) | 79 | 69 | 73
Pharyngitis (Infections and infestations) | 13 | 16 | 16
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 12 | 7
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 18 | 8 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No